CLINICAL TRIAL: NCT06086002
Title: Evaluation of Clinical Feasibility of Microwave Ablation Using Two Channel Microwave Generator and Two Antennas for Small Hepatocellular Carcinoma: A Preliminary Prospective Single Center Study
Brief Title: Clinical Feasibility of Microwave Ablation Using Two Channel Microwave Generator and Two Antennas for Small Hepatocellular Carcinoma
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Jeong Min Lee, Professor, Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2308-023-1457
Record Dates: First submitted 2023-10-10; First posted 2023-10-17 (Actual); Last update posted 2023-10-17 (Actual); Status verified 2023-10

CONDITIONS: Hepatocellular Carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Overlapping ablation with single antenna (Active Comparator)
  Interventions: Device: Microwave ablation
- Simultaneous ablation with two antennas (Experimental)
  Interventions: Device: Microwave ablation

INTERVENTIONS:
Device: Microwave ablation — Microwave ablation will be performed by using single antenna (Emprint, Medtronic) with overlapping ablation or two antennas (Starwave, STARmed) with simultaneous ablation.

SUMMARY:
To compare safety and efficacy of microwave ablation with simultaneous ablation using two antennas versus overlapping ablation with single antenna for small hepatocellular carcinoma

ELIGIBILITY:
Inclusion Criteria:

* Child-Pugh Class A or B
* chronic hepatitis B or chronic hepatitis C or liver cirrhosis
* presence of hepatocellular carcinoma (HCC) confirmed by pathology or imaging studies including contrast enhanced computed tomography (CT) or magnetic resonance imaging (MRI) according to Liver Imaging Reporting and Data System (LI-RADS) v2018
* single lesion less than or equal to 3 cm, or up to 3 lesions, each greater than less than or equal to 3 cm at the time of locoregional treatment

Exclusion Criteria:

* number of recurrent HCCs, equal or more than 3
* largest recurrent HCC size over 3 cm
* presence of vascular invasion by HCC
* diffuse infiltrative type HCC
* HCCs located less than 5 mm from central bile duct or large portal vein or large hepatic vein
* platelet count less than 40,000 per mm3 or International Normalized Ratio (INR) prolongation over 50%
* presence of extrahepatic metastasis

Ages: 20 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2023-09-18 (Actual); Primary Completion 2024-10 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Technical success | Immediately after ablation
  Evaluate technical success defined as complete ablation of the index tumor with safety margin, equal or larger than 5 mm on immediate CT.
Technique efficacy | 1 month after ablation
  Evaluate technical success defined as complete ablation of the index tumor on 1 month follow-up CT.

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National University Hospital, Seoul, South Korea